CLINICAL TRIAL: NCT06395051
Title: Acute Effects of Ketone Monoester Supplementation on Brain Function in Older Men with Overweight
Brief Title: Effects of Ketone Monoesters on Brain Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: METC24-008
Record Dates: First submitted 2024-04-29; First posted 2024-05-01 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Brain Insulin Sensitivity; Brain Vascular Function; Cerebral Blood Flow; Cognitive Performance; Appetite Control

STUDY DESIGN:
Intervention Model Description: Study participants will receive in random order acutely 395 mg/kg body weight ketone monoesters or placebo, seperated by a wash-out period of at least 1 week.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental (Experimental): Ketone monoesters
  Interventions: Dietary Supplement: Ketone Monoester
- Placebo (Placebo Comparator): Taste- and volume-matched placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone Monoester — Ketone monoester supplement (395 mg/kg body mass)
  Arms: Experimental
Dietary Supplement: Placebo — The placebo will be taste-matched to the active supplement for bitterness using denatonium benzoate and volume-matched with water
  Arms: Placebo

SUMMARY:
Disturbances in brain insulin-sensitivity are not only observed in obesity and type 2 diabetes (T2D), but also during brain aging and in dementia. Ketone monoester supplements may improve brain insulin-sensitivity, which can be quantified by measuring the gray-matter cerebral blood flow (CBF) response to intranasally administered insulin. We hypothesize that acute ketone monoester supplementation increases (regional) brain vascular function and insulin-sensitivity thereby improving cognitive performance and appetite control. The primary objective is to evaluate in older men the acute effect of ketone monoester supplementation on (regional) brain vascular function and insulin-sensitivity, as quantified by the non-invasive gold standard magnetic resonance imaging (MRI)-perfusion method Arterial Spin Labelling (ASL). The CBF response to intranasal insulin is a robust and sensitive physiological marker of brain insulin-sensitivity. Secondary objectives are to investigate effects on cognitive performance as assessed with a neuropsychological test battery, and appetite control as quantified by functional MRI (fMRI) with visual food cues.

ELIGIBILITY:
Inclusion Criteria:

* Men, aged between 60-75 years
* BMI between 25-30 kg/m2
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum TC < 8.0 mmol/L
* Fasting serum TAG < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Women
* Left-handedness
* Following a low-carbohydrate diet or consuming nutritional ketone supplements
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of products or dietary supplements known to interfere with the main outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid or glucose metabolism, or neurological or mental disorders.
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g. pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia).

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2024-07-03 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-11-15 (Actual)

PRIMARY OUTCOMES:
Brain Vascular Function | Change from placebo intervention at 30 minutes after supplement intake
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)
Brain Insulin Sensitivity | Change from placebo intervention at 60 minutes after supplement intake
  Cerebral blood flow measurements before and after a nasal insulin spray as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Appetite-related brain reward activity | Change from placebo intervention at 40 minutes after supplement intake
  Blood oxygenation level-dependent (BOLD)-functional MRI (fMRI) response to food cues
Cognitive Performance | Change from placebo intervention at 120 minutes after supplement intake
  Cambridge Neuropsychological Test Automated Battery (CANTAB)
Brain Perfusion | Change from placebo intervention at 120 minutes after supplement intake
  Transcranial Doppler (TCD) ultrasound will be used to assess the velocity of blood flow through the middle cerebral artery (MCA)
Blood pressure | Change from placebo intervention at 90 minutes after supplement intake
  Office blood pressure and heart rate
Ketone metabolism | During 120 minutes following supplement intake
  Circulating beta-hydroxybutyrate concentrations
Glucose metabolism | During 120 minutes following supplement intake
  Circulating glucose and insulin concentrations
Markers related to low-grade systemic inflammation | During 120 minutes following supplement intake
  Circulating high-sensitive C-reactive protein concentrations
Appetite hormones | During 120 minutes following supplement intake
  Circulating ghrelin concentrations
Perceived hunger and satiety | During 120 minutes following supplement intake
  Visual analogue scale (VAS) questionnaires
Anthropometric measurements | Before supplement intake
  Weight, length, waist and hip circumference
Food intake | Once 120 minutes following supplement intake
  Food Frequency Questionnaire to assess food intake over the past month

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No